CLINICAL TRIAL: NCT01592799
Title: Burden of Influenza-related Hospitalizations and Emergency Room Visits in Children in Spain
Brief Title: Study on the Burden of Influenza-related Hospitalizations and Emergency Room (ER) Visits in Children in Spain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 114004
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-06

CONDITIONS: Influenza
Keywords: Influenza; Children; Hospitalizations; Spain; Burden
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

ARMS (1):
- Influenza Group (Other): Children <15 years of age hospitalized for or presenting to an ER for acute ARI and/or isolated fever during the influenza season.
  Interventions: Procedure: Throat swab and/or nasopharyngeal swab; Other: Data collection

INTERVENTIONS:
Procedure: Throat swab and/or nasopharyngeal swab — Samples will be tested to quantify the inpatient and ER visits burden of laboratory-confirmed influenza.
Other: Data collection — Log Sheet will be used to collected data on a monthly basis for the following age groups: < 6 months; 6-23 months; 24-59 months; > 5 years.

SUMMARY:
This study aims to quantify the inpatient and ER visits burden of laboratory-confirmed influenza, and compare the clinical features, severity, complications, risk factors and socioeconomic impact of influenza in children presenting with acute respiratory illness (ARI) and/or isolated fever, with or without laboratory-confirmed influenza.

DETAILED DESCRIPTION:
The total medical cost associated with each hospitalization or ER visit will also be calculated at the end of this study.

The study will be conducted from October, 2010, until May, 2011. Each subject will be followed-up for 21-30 days via telephone. The follow-up medical chart review will preferably be performed within 7 days after the telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom the investigator believes that they and/or their parents/guardians can and will comply with the requirements of the protocol.
* A male or female <15 years of age at the time of study entry. A subject will become ineligible on his/her 15th birthday.
* Signed informed consent from the parents or guardians of the subject and signed assent from children ≥ 12 years old.
* Presenting with a sudden onset clinical process comprising :

  * Isolated fever defined as: oral temperature ≥ 37.5°C / axillary temperature ≥ 37.5°C / Rectal temperature ≥ 38°C / tympanic temperature on oral setting ≥ 37.5°C / tympanic temperature on rectal setting ≥ 38°C without an obvious cause.

And/or

* ARI defined as one or more of the following symptoms: sore throat, coryza, cough, breathing difficulties.

Exclusion Criteria:

• Children in foster care.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 501 (Actual)
Dates: Start 2010-11-23; Primary Completion 2011-05-23 (Actual); Study Completion 2011-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bilbao, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in October, 2010, and last until May, 2011, or until the target sample size was enrolled.
Groups:
- Influenza Group: Children <15 years of age hospitalized for or presenting to an Emergency Room (ER) for Acute Respiratory Illness (ARI) and/or isolated fever during the influenza season.
Period: Overall Study
Arm/Group | Influenza Group
Started | 501
Completed | 501
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Influenza Group: Children less than (<) 15 years of age hospitalized for or presenting to an ER for acute ARI and/or isolated fever during the influenza season.
Arm/Group | Influenza Group
Number analyzed (Participants) | 501
Age, Continuous [Mean (Standard Deviation); unit: Months] | 33.0 (37.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212
  Male | 289

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Laboratory-confirmed Influenza Presenting With an Acute Respiratory Illness (ARI) and/or Isolated Fever
Description: ARI was defined as one or more of the following symptoms: sore throat (in children greater than or equal to (≥) 3 years old), coryza (runny nose), cough, breathing difficulties. Isolated fever was defined as: oral temperature ≥37.5°C / axillary temperature ≥37.5°C / Rectal temperature ≥38°C / tympanic temperature on oral setting ≥37.5°C / tympanic temperature on rectal setting ≥38°C without an obvious cause.
Time Frame: Day 0 till Day 28-37
Population: The analysis was performed on the according-to-protocol (ATP) cohort for analysis, which included all evaluable subjects (i.e. those meeting all eligibility criteria and complying with the procedures defined in the protocol) for whom data concerning endpoint measures were available.
Measure: Count of Participants; unit: Participants
Groups:
- Influenza Group: Children <15 years of age hospitalized for or presenting to an ER for ARI and/or isolated fever during the influenza season.
Arm/Group | Influenza Group
Number analyzed (Participants) | 501
Participants
  Emergency Room | 120
  Hospitalized | 11

2. Primary Outcome: Direct Medical Cost Per Hospitalization or ER Visit With Laboratory-confirmed Influenza
Description: Ward specific room charge and Intensive Care Unit (ICU) were computed as daily charge multiplied by the number of days.
Time Frame: Day 0 till Day 28-37
Population: The analysis was performed on the according-to-protocol (ATP) cohort for analysis, which included all evaluable subjects (i.e. those meeting all eligibility criteria and complying with the procedures defined in the protocol) for whom data concerning endpoint measures were available and who were hospitalized or visited an emergency room.
Measure: Mean (Standard Deviation); unit: Euros
Arm/Group | Influenza Group
Number analyzed (Participants) | 131
Euros
  Laboratory | 57.27 (48.93)
  Radiology | 16.94 (9.68)
  Other diagnostics | 89.94 (80.25)
  Total for diagnostics | 52.97 (63.77)
  Prescribed medication [given in the hospital] | 5.52 (10.25)
  Prescribed medication | 12.28 (18.49)
  Non-prescribed medication | 9.86 (12.56)
  Total for treatments | 16.44 (21.68)
  Ward specific room charge | 1774.55 (1062.94)
  ICU | 1535.19 (0.0)
  Total for inpatient charge | 1884.21 (1182.22)
  ER visit | 170.16 (64.18)
  Others | 136.77 (49.91)

3. Secondary Outcome: Number of Subjects With Other Laboratory-confirmed Respiratory Viruses
Description: Among the other laboratory-confirmed respiratory viruses there were:adenovirus, respiratory syncytial virus, parainfluenza virus 1, 2 and 3, metapneumovirus, bocavirus, rhinovirus or coronavirus. The outcome was assessed in subjects with an acute respiratory illness (ARI) and/or isolated fever episode.
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Group
Number analyzed (Participants) | 501
Participants
  Emergency Room | 98
  Hospitalized | 47

4. Secondary Outcome: Number of Subjects With Fatal Outcomes
Description: Deaths from ARI and/or fever episodes by laboratory-confirmed influenza status were assessed.
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Influenza Positive Group: Children <15 years of age with at least one laboratory test positive for influenza.
- Influenza Negative Group: Children <15 years of age with no laboratory test positive for influenza.
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Participants | 0 | 0

5. Secondary Outcome: Number of Subjects With Secondary Bacterial Infections
Description: The outcome assessed the various complications by laboratory-confirmed influenza status.
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Participants
  Any complication | 37 | 145
  Secondary bacterial pneumonia | 11 | 34
  Primary influenza viral pneumonia | 3 | 7
  Bronchiolitis | 10 | 67
  Acute Otitis Media | 12 | 33
  Myositis | 2 | 1
  Pericarditis | 0 | 0
  Conjunctivitis | 3 | 16

6. Secondary Outcome: Number of Subjects With Potential Risk Factors at Study Start by Laboratory-confirmed Influenza Status
Description: Risk factors were classified as pre-existing conditions, breast-feeding status and day-care status.
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Participants
  Any pre-existing conditions | 32 | 82
  No pre-existing conditions | 99 | 288
  Prematurity (<36 weeks gestation) | 1 | 12
  Chronic pneumopathy (including asthma) | 25 | 60
  Cardiovascular disease | 1 | 2
  Neuromuscular diseases | 0 | 1
  Other | 7 | 15
  Breast fed | 15 | 88
  Not breast fed | 35 | 153
  Breast feeding status not known (>2 years old) | 81 | 129
  In day-care attendance | 60 | 176
  Not in day-care attendance | 28 | 152
  Not known if in day-care attendance (>5 years old) | 43 | 42

7. Secondary Outcome: Number of Days of Hospitalization
Description: The outcomes was assessed in subjects with laboratory-confirmed influenza status
Time Frame: Day 0 till Day 28-37 (between October 2010 until May 2011)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Days | 2.0 (0.00) | 4.4 (4.34)

8. Secondary Outcome: Number of Subjects Using Any ARI and/or Fever Related Medication Taken Prior to Hospitalization or ER Visit by Laboratory-confirmed Influenza Status
Description: ARI and/or fever related medication included: antivirals, antibiotics, cough suppressants, pain medication, antipyretics and mucolytics.
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Participants
  Any medication | 119 | 300
  Antibiotics | 9 | 21
  Cough suppressants | 3 | 7
  Antihistamines | 1 | 1
  Pain medication | 12 | 21
  Antipyretics | 114 | 267
  Mucolytics | 1 | 5
  Other medication | 10 | 61

9. Secondary Outcome: Number of Subjects Using Any ARI and/or Fever Related Medication Prescribed During Hospitalization or ER Visit by Laboratory-confirmed Influenza Status
Description: as for outcome 8
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Participants
  Any medication prescribed | 122 | 344
  Antivirals | 4 | 1
  Antibiotics | 17 | 77
  Cough suppressants | 1 | 0
  Pain medication | 12 | 28
  Antipyretics | 120 | 284
  Mucolytics | 0 | 1
  Other medication | 17 | 114

10. Secondary Outcome: Number of Subjects Using Any ARI and/or Fever Related Medication Prescribed Since Hospitalization or ER Visit by Laboratory-confirmed Influenza Status
Description: as for outcome 8
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Participants
  Any medication prescribed | 130 | 367
  Antivirals | 3 | 0
  Antibiotics | 41 | 151
  Cough suppressants | 6 | 3
  Antihistamines | 0 | 4
  Pain medication | 7 | 18
  Antipyretics | 121 | 287
  Mucolytics | 3 | 9
  Other medication | 35 | 162

11. Secondary Outcome: Number of Subjects Using Any Non-prescribed ARI and/or Fever Related Medication Taken Since Hospitalization or ER Visit
Description: as for outcome 8
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Participants
  Any non-prescribed medication | 9 | 30
  Antibiotics | 2 | 11
  Antihistamines | 0 | 1
  Pain medication | 1 | 3
  Antipyretics | 0 | 2
  Mucolytics | 0 | 1
  Other medication | 6 | 16

12. Secondary Outcome: Number of Days of School Absenteeism
Description: School absenteeism was assessed among patients during the follow-up period by laboratory-confirmed influenza status.
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Days | 6.6 (3.46) | 6.4 (3.66)

13. Secondary Outcome: Number of Days of Parent or Caregiver Time Off Work
Description: This outcome assessed absenteeism among caregivers to provide patient care during the follow-up period by laboratory-confirmed influenza status.
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Days | 4.4 (2.76) | 4.1 (3.10)

14. Secondary Outcome: Number of Subjects With Household Members With Influenza-like Illness
Description: This outcome assessed the number of cases with household contacts presenting influenza like illness symptoms during the follow-up period by laboratory-confirmed influenza status.
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Number; unit: Household members
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Household members
  Household members with influenza-like illness | 73 | 146
  Household members with no influenza-like illness | 58 | 224
  1-2 household members with ARI/fever | 19 | 35
  3-4 household members with ARI/fever | 48 | 98
  >4 household members with ARI/fever | 6 | 12
  Missing confirmed | 0 | 1

15. Secondary Outcome: Proportion of Household Members Presenting Influenza Like Illness Symptoms (ARI and/or Isolated Fever)
Description: This outcome assessed the proportion of influenza like illness (ILI) among household members of children < 15 years with and without laboratory-confirmed influenza.
Time Frame: Day 0 till Day 28-37
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of household members
Arm/Group | Influenza Positive Group | Influenza Negative Group
Number analyzed (Participants) | 131 | 370
Percentage of household members | 25.80 [21.16 to 31.06] | 17.45 [15.02 to 20.18]

ADVERSE EVENTS:
Time Frame: No solicited or unsolicited adverse events were collected during this study. No SAEs or fatal events were recorded during this study.
Description: Serious and non-serious adverse events were not planned to be assessed as part of this study protocol.
Arm/Group | Influenza Group
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.